CLINICAL TRIAL: NCT02213965
Title: Clinical Investigation Acc. to MPG §23b: Open-label Prospective Study Comparing the Handling of the Handling of Two Peripheral IV Catheter (PIV) Systems (Ported and Non Ported) in Randomized Order
Brief Title: Study Comparing the Handling of Two Peripheral IV Catheter Systems
Status: Completed | Type: Observational
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Other Study IDs: HC-O-H 1411
Record Dates: First submitted 2014-07-22; First posted 2014-08-12 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Intravenous Access According to Instructions For Use
Keywords: Intravenous Catheter; Vasofix safety; Introcan safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vasofix® Safety: Peripheral IV catheter Vasofix® Safety
  Interventions: Device: Peripheral IV catheter
- Introcan Safety®: Peripheral IV catheter Introcan Safety® IV catheter
  Interventions: Device: Peripheral IV catheter

INTERVENTIONS:
Device: Peripheral IV catheter — Intravenous access according to Instructions For Use

SUMMARY:
A peripheral intravenous catheter is the most commonly used vascular access device in medicine. Primary objective is to compare insertion and handling of two peripheral intravenous catheters in clinical routine.

ELIGIBILITY:
Inclusion:

* Patients of the center Anesthesiology, Operating-Room Management and Intensive Care Medicine, Gynaecology and Paediatrics in need for peripheral intravenous access
* Male and female patients, adult and paediatric
* Is able to give written informed consent, for children the legal representatives

Exclusion:

* Participation in another intervention trial during the study
* Lacking willingness to save and hand out data within the study
* Accommodation in an institution due to an official or judicial order
* The potential insertion site shows deformities, phlebitis, infiltration, dermatitis, burns, lesions, nerve injuries with paresthesia or tattoos
* Study PIV catheter site will be placed below an old infusion site
* Patient has a documented or known allergy sensitivity to a medical adhesive product such as transparent film, adhesive dressing, tapes or liquid skin protectants
* Patient requires the application of a topical ointment, or solution under the dressing in addition to the prep required in the protocol
* Patient has or had previous IV catheter-related phlebitis or infiltration during this hospitalization
* Patients with fear of injection
* Preterm infants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children
Sampling Method: Probability Sample
Enrollment: 2340 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Incidence of successful puncturing on the first attempt | From catheter fixation until the stay in operation theatre and/or recovery room up to 12 hours

SECONDARY OUTCOMES:
Rate of insertion failures | From catheter fixation until the stay in operation theatre and/or recovery room up to 12 hours
Rate of difficulties to insert catheter and to withdraw the needle with regard to:Penetration characteristics of the needle, insertion and movement of catheter | From catheter fixation until the stay in operation theatre and/or recovery room up to 12 hours
Rate and number of testing of ease of moving | From catheter fixation until the stay in operation theatre and/or recovery room up to 12 hours
Rate and number of recannulation | From catheter fixation until the stay in operation theatre and/or recovery room up to 12 hours
Rate, number and kind/extend of blood emission | From catheter fixation until the stay in operation theatre and/or recovery room up to 12 hours
Incidence of needle stick injuries | During catheter fixation
Condition of fixation after completion of catheter insertion | During catheter fixation until directly after catheter insertion
  dry and clean, moisturized, soiled?
Rate of adherence to standard application requirements of catheter placement | During catheter fixation until directly after catheter fixation
For Vasofix Safety: Rate and nature of use of application port | From catheter fixation until the stay in operation theatre and/or recovery room up to 12 hours
General judgment of catheter (school class grading) | From catheter fixation until the stay in operation theatre and/or recovery room up to 12 hours
Adverse Events | From catheter fixation until the stay in operation theatre and/or recovery room up to 12 hours

OTHER OUTCOMES:
Age and gender of the patient | At the beginning of the investigation
ASA score of the patient | At the beginning of the investigation
Weight and height of the patient | At the beginning of the investigation
Vein and skin condition of the patient | At the beginning of the investigation
Location of Peripheral Intervenous Catheter | After catheter fixation
Judgment on application port and wings given by user | From catheter fixation until the stay in operation theatre and/or recovery room up to 12 hours
Working experience of the user | At the beginning of the investigation
  Working experience of the user in a hospital in at the beginning of the investigation
Function of the user | At the beginning of the investigation
  Job title of the user

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, Univ.- Prof. Dr., Principal Investigator — Klinik für Anästhesiologie mit Schwerpunkt operative Intensivmedizin CVK/CCM, Charité-Universitätsmedizin Berlin
Locations (2):
- Germany (2):
  - Klinik für Anästhesiologie mit Schwerpunkt operative Intensivmedizin CVK/CCM, Charité-Universitätsmedizin Berlin, Berlin
  - Universitätsklinik für Anästhesiologie und Intensivmedizin Tübingen, Tübingen

REFERENCES:
- [Derived] Morgeli R, Schmidt K, Neumann T, Kruppa J, Fohring U, Hofmann P, Rosenberger P, Falk E, Boemke W, Spies C. A comparison of first-attempt cannulation success of peripheral venous catheter systems with and without wings and injection ports in surgical patients-a randomized trial. BMC Anesthesiol. 2022 Mar 31;22(1):88. doi: 10.1186/s12871-022-01631-7. PMID 35361115